CLINICAL TRIAL: NCT05809648
Title: A Prospective, Blinded, Observational Study to Assess the Accuracy of Magnetocardiography (MCG) as a Tool for Diagnosing Acute Coronary Syndrome (ACS) in Emergency Department Patients Presenting With Acute Chest Pain
Brief Title: A Study to Assess the Accuracy of Magnetocardiography (MCG) to Diagnose True Ischemia in Patients With Chest Pain in the ED
Acronym: MCG
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sara A. Hevesi, Principal Investigator, Mayo Clinic
Other Study IDs: 20-001225
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Chest Pain; Emergency Medicine
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of the research is to see if patients that come to the Emergency Department with chest pain can be more accurately and more quickly diagnosed by magnetocardiography (MCG) to see if their chest pain is caused by coronary ischemia (reduced blood flow to the heart) in patients with normal or have non-specific changes on the ECG vs other causes by other reasons.

DETAILED DESCRIPTION:
Hypothesis: MCG can accurately, and in real-time, identify an acute coronary syndrome for patients presenting to the emergency department (ED) with chest pain and is faster than current practice.

Aims, purpose, or objectives: Our primary objective is to measure the diagnostic accuracy of the Mesuron Avalon-H90 MCG device to detect ACS (unstable angina, NSTEMI) in Emergency Department patients who present with acute chest pain when compared to the current goal standard.

Our secondary objectives are as follows:

* To study the ability of MCG to rule in or rule out ACS in real-time. We will assess the value of the MCG results in conjunction with the HEART pathway score. This will include looking at the diagnostic test accuracy, sensitivity and specificity of the device when used in conjunction with and without the HEART Pathway score, including versus excluding the troponin level (as the results of this is usually delayed by 45 minutes to 1 hour). In this way, we hope to demonstrate this technology may decrease ED length of stay in chest pain patients and decrease time to diagnosis. The comparison goal standard will be the Cardiology diagnosis, the result of serial troponins, or the ED diagnosis depending on the disposition of the patient.
* To estimate ability of MCG for prognostication for major adverse cardiac events (MACE) at 3 days, 7 days, 30 days and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the ED with acute chest pain when an ACS is on the differential diagnosis.
* Patient willing and able to give informed consent.

Exclusion Criteria:

* ST elevation > 1 mm on any two contiguous ECG leads.
* Hemodynamic instability (SBP >220 or <80, HR >160).
* Pregnant patients.
* Incarcerated patients (FMC patients).
* Patients with a pacemaker or defibrillator.
* Metal implants in the body (that are not MRI safe).
* Patients that are unable to lie down in the MCG machine or stay still.
* Patients who are unable to understand the informed consent process (ex: non-English speakers without an available interpreter, cognitive delay).
* Patients without the capacity to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting with chest pain to the Mayo Clinic Minnesota, Saint Mary's hospital emergency department (ED).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy | 12 months
  Our primary objective is to measure the diagnostic accuracy of the Mesuron Avalon-H90 MCG device to detect ACS (unstable angina, NSTEMI) in Emergency Department patients who present with acute chest pain when compared to the current goal standard.

SECONDARY OUTCOMES:
Real-time rule out of ACS | 12 months
  • To study the ability of MCG to rule in or rule out ACS in real-time. We will assess the value of the MCG results in conjunction with the HEART pathway score. This will include looking at the diagnostic test accuracy, sensitivity and specificity of the device when used in conjunction with and without the HEART Pathway score, including versus excluding the troponin level (as the results of this is usually delayed by 45 minutes to 1 hour). In this way, we hope to demonstrate this technology may decrease ED length of stay in chest pain patients and decrease time to diagnosis. The comparison goal standard will be the Cardiology diagnosis, the result of serial troponins, or the ED diagnosis depending on the disposition of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Hevesi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials